CLINICAL TRIAL: NCT06975488
Title: Comparison Between Fragmentation and Dusting Modalities Utilizing Holmium YAG Laser in Ureteroscopy for Ureteral Stone Treatment
Brief Title: Effectiveness of LASER in Treatment of Ureteric Stones.
Acronym: LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: District Headquarters Teaching Hospital Sahiwal (Other)
Responsible Party: Principal Investigator, Ussama Iftikhar, Resident, District Headquarters Teaching Hospital Sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 195
Record Dates: First submitted 2025-05-03; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ureteric Stone
Keywords: Laser; URS; DJ Stent; Lithotripsy; ESWL; URSL
MeSH Terms: conditions — Ureterolithiasis | interventions — Lithotripsy, Laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A patients will be treated with fragmentation modality utilizing Holmium YAG laser.
  Interventions: Procedure: LASER Lithotripsy ( Fragmentation modality)
- Group B (Experimental): Group B patients will be treated with dusting modality utilizing Holmium YAG laser.
  Interventions: Procedure: LASER lithotripsy (Dusting Modality)

INTERVENTIONS:
Procedure: LASER Lithotripsy ( Fragmentation modality) — Group-A patients will be treated with fragmentation modality utilizing Holmium YAG laser.
  Arms: Group A
Procedure: LASER lithotripsy (Dusting Modality) — Group-B patients will be treated with dusting modality utilizing Holmium YAG laser.
  Arms: Group B

SUMMARY:
Ureteroscopic laser lithotripsy is becoming the most commonly utilized treatment for patients with ureteral stone. The Holmium: YAG laser is integral to the operation and is the preferred flexible intracorporeal lithotripsy. It is considered cost-effective and efficient choice in ureteroscopic lithotripsy on all types of stones. As in recent years, there has been increasing interest in examining the effect of varying the laser settings on the effectiveness of stone treatment. The objective of the study is to compare the fragmentation and dusting modalities utilizing Holmium YAG laser in ureteroscopy for ureteral stone treatment. It will be a randomized control trial (RCT) in which 160 patients visiting Sahiwal Teaching Hospital, Sahiwal will be included. The patients will be divided into two groups. Group-A patients will be treated with fragmentation modality utilizing Holmium YAG laser while Group-B patients will be treated with dusting modality utilizing Holmium YAG laser. Simple random sampling technique will be carried out. The patients' age, gender, stone number, stone laterality, stone location, ureteral condition, reteropulsion, stricture formation, stone clearance, operative time, hospital stay, presence of retropulsion and complications will be recorded. Data will be collected through proforma, which will be entered and analyzed using SPSS version 26.0. For quantitative variables such as: age, operation time, hospital stay, stone number ,mean and standard deviation will be calculated and for qualitative variables such as: gender, and laterality, stone location, ureter condition, prevalence of pyuria, stone clearance, presence of retropulsion, ureter injury, frequency and percentages will be calculated. Data will be presented in tables and graphs for both quantitative and qualitative variables. Chi-square test will be used to estimate the association between study variables. P-value <0.05 will be considered significant. It is anticipated that the results of this study will be helpful for health care planners and surgeons to provide better treatment option to the patients with ureteral stone.

ELIGIBILITY:
Inclusion Criteria:

1. Stone size 1cm to 1.5cm at proximal Ureter.
2. Patients aged between 15 to 70 years.
3. Both genders.

Exclusion Criteria:

1. Patients with active urinary tract infection
2. Pregnancy
3. Immunocompromised patients

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Stone Free Rate | There would be 4 follow up visits. First visit will be after 1 week of URSL and X Ray KUB will be done. Second visit will be after 2 weeks of URSL and we will plan the removal of DJ stent. Those cases in which ureteral inury is suspected or stone burden
  Stone-free will be defined as no residual stones > 3 mm in the ureter of the affected side at one month postoperatively on computerized tomography (CT KUB Plain).
Reteropulstion | During procedure.
  Retropulsion, defined as unintended migration of stone into the kidney, leads to failure and results in a lower SFR.

SECONDARY OUTCOMES:
Uretral Stricture Formation | Post-URS ureteral stricture is defined as complete or partial ureteral obstruction as shown by the excretory phase of CTU, which was confirmed with delayed or absent radioactive tracer washout at 8 weeks after stent removal.
  Post-URS ureteral stricture is defined as complete or partial ureteral obstruction as shown by the excretory phase of CTU, which was confirmed with delayed or absent radioactive tracer washout at 8 weeks after stent removal.

CONTACTS AND LOCATIONS:
Overall Officials: U A IFTIHKAR, MS, Principal Investigator — District Headquarters Teaching Hospital Sahiwal; A RIAZ, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- District Headquarters Teaching Hospital Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen BH, Lin TF, Tsai CC, Chen M, Chiu AW. Comparison of Fragmentation and Dusting Modality Using Holmium YAG Laser during Ureteroscopy for the Treatment of Ureteral Stone: A Single-Center's Experience. J Clin Med. 2022 Jul 17;11(14):4155. doi: 10.3390/jcm11144155. PMID 35887919
- See also: Laser lithotripsy in treatment of ureteric stones — https://pmc.ncbi.nlm.nih.gov/articles/PMC9324266/